CLINICAL TRIAL: NCT03583775
Title: Comprehensive Free-breathing 3D Cine Cardiovascular Magnetic Resonance
Brief Title: 3D Cine Cardiovascular Magnetic Resonance
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Andrew Powell, Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: IRB-P00028262
Record Dates: First submitted 2018-06-27; First posted 2018-07-11 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with congenital heart disease: Patients with congenital heart disease who are greater than 40 kg and are referred for a clinically indicated 2D CMR exam with a gadolinium-based contrast agent.
  Interventions: Other: Cardiovascular Magnetic Resonance Imaging

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance Imaging — Cardiovascular Magnetic Resonance Imaging or MRI exam from children's with congenital heart disease

SUMMARY:
Conventional CMR is based on breath-hold 2D cine image acquisitions which are sequentially acquired in different imaging planes. The necessity of precisely planning and then acquiring multiple 2D imaging planes during breath-hold is relatively inefficient and leads to CMR exam times of ≤60 minutes. However, some patients are too ill or young to hold their breath. Furthermore, 2D images sometimes fail to provide a complete picture of complex 3D anatomy of patients with complex morphology.

To address these limitations, we have recently developed a 3D cine (3 spatial dimensions plus time) CMR technique. Rather than acquiring 2D cine images in multiple orientations during breath-hold, this approach allows one to acquire a free-breathing 3D block of data for each phase of cardiac cycle that can be reformatted offline into the desired views without adding to the exam time. This added efficiency should lead to a reduction in CMR exam time, increasing patient comfort, and making CMR exam easy and available for all. In addition, the 3D nature of the data may yield more complete information about the anatomy and physiology.

In this proposal, we will examine the agreement between the 2D cine and 3D cine CMR techniques with regard to left and right ventricular volumes and systemic and pulmonary blood flow circulation. The internal consistency of the measurements between the 2 techniques will be also investigated. This study will focus on children because they may benefit the most from the short, improved efficiency, and free-breathing CMR exams.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are greater than 40 kg and are referred for a clinically indicated 2D CMR exam with a gadolinium-based contrast agent. Informed consent/assent will be obtained.

Exclusion Criteria:

* Patients who are under anesthesia, sedated, or with a contraindication to CMR exams.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with different races and ethnicity are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
End-diastolic and end-systolic volumes of right and left ventricles | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Tarek Alsaied, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided